CLINICAL TRIAL: NCT00467025
Title: A Randomized, Double Blinded, Multi-Center Phase 2 Study to Estimate the Efficacy and Evaluate the Safety and Tolerability of Sorafenib in Combination With AMG 386 or Placebo In Subjects With Metastatic Clear Cell Carcinoma of the Kidney
Brief Title: AMG 386, 20060159 Phase 2, RCC 1st Line in Combination With Sorafenib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060159
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Advanced Renal Cell Carcinoma
Keywords: Metastatic clear cell carcinoma of the kidney; RCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — trebananib; Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental)
  Interventions: Drug: AMG 386; Drug: Sorafenib; Drug: AMG 386 placebo IV
- Arm B (Experimental)
  Interventions: Drug: AMG 386; Drug: Sorafenib
- Arm C (Active Comparator)
  Interventions: Drug: Sorafenib; Drug: AMG 386 placebo IV

INTERVENTIONS:
Drug: AMG 386 — 3 mg/kg or 10mg/kg IV weekly until unacceptable toxicity or disease progression
  Arms: Arm A; Arm B
Drug: Sorafenib — 400 mg PO BID
Drug: AMG 386 placebo IV — AMG 386 placebo IV
  Arms: Arm A; Arm C

SUMMARY:
This is a phase 2, randomized, double-blind, placebo controlled, multi-center study to estimate the improvement in progression free survival (PFS) and evaluate the safety and tolerability of AMG 386 in combination with sorafenib in the treatment of subjects with advanced clear cell carcinoma of the kidney.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologically confirmed metastatic RCC with a clear cell component
* Low or intermediate risk according to the Memorial Sloan Kettering Cancer Center (MSKCC) prognostic risk classification.
* Measurable disease with at least one unidimensionally measurable lesion per RECIST guidelines with modifications
* Adequate organ and hematological function as evidenced by laboratory studies conducted at Screening.
* ECOG of 0 or 1

Exclusion Criteria:

Disease Related

* Known history of central nervous system metastases.
* Previous treatment (excluding surgery and palliative radiotherapy) for advanced or metastatic renal cell carcinoma
* Focal radiation therapy for palliation of pain from bony metastases within 14 days of randomization.

Medications

* Currently or previously treated with inhibitors of VEGF.
* Currently or previously treated with inhibitors of angiopoietin or Tie2.
* Currently or previously treated with bevacizumab.

General Medical

* Diagnosis of acute pancreatitis.
* Myocardial infarction, cerebrovascular accident, transient ischemic attack, percutaneous transluminal coronary angioplasty/stent, congestive heart failure, grade 2 or greater peripheral vascular disease, arrhythmias not controlled by outpatient medication, or unstable angina within 1 year prior to randomization
* Major surgery within 30 days before randomization or still recovering from prior surgery
* Uncontrolled hypertension as defined as diastolic > 90 mmHg OR systolic >150 mmHg. Anti-hypertensive medications are permitted.

Other

* Other investigational procedures are excluded
* Subject currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s), or subject is receiving other investigational agent(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2007-05; Primary Completion 2010-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 2 3/4 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 3/4 years
Duration of response (DOR) | 2 3/4 years
Change in continuous measures of tumor burden | 2 3/4 years
Time-adjusted area under the curve (AUC) for the FACT-Kidney Cancer Symptom Index (FKSI-15) scale score from baseline through disease progression with imputation for missing data | 2 3/4 years
Incidence of AEs and significant laboratory changes | 2 3/4 years
Incidence of the occurrence of anti-AMG 386 antibody formation | 2 3/4 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Rini B, Szczylik C, Tannir NM, Koralewski P, Tomczak P, Deptala A, Dirix LY, Fishman M, Ramlau R, Ravaud A, Rogowski W, Kracht K, Sun YN, Bass MB, Puhlmann M, Escudier B. AMG 386 in combination with sorafenib in patients with metastatic clear cell carcinoma of the kidney: a randomized, double-blind, placebo-controlled, phase 2 study. Cancer. 2012 Dec 15;118(24):6152-61. doi: 10.1002/cncr.27632. Epub 2012 Jun 12. PMID 22692704
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com